CLINICAL TRIAL: NCT06941610
Title: An Evaluation of the Erchonia Corporation GVS Laser As a Non-Invasive Treatment to Improve the Appearance of Skin Laxity on the Abdominal Region
Brief Title: An Evaluation of the Erchonia Laser As a Non-Invasive Treatment to Improve the Appearance of Skin Laxity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-LAX
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Erchonia GVS Laser (Experimental): 405nm violet and 520nm green laser light therapy.
  Interventions: Device: Erchonia GVS Laser

INTERVENTIONS:
Device: Erchonia GVS Laser — 405nm violet and 520nm green laser light therapy.

SUMMARY:
The purpose of this clinical study is to determine the effectiveness of the Erchonia® GVS in improving the appearance of skin laxity on the abdominal region.

DETAILED DESCRIPTION:
This clinical study is a prospective open-label design with post-study independent blinded outcome analysis to evaluate the efficacy of the Erchonia® GVS Laser in improving the appearance of skin laxity on the abdominal region. Participants will receive 8 treatments over the course of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed a written informed consent form.
* Male or female 22 to 70 years of age, inclusive.
* Desire to undergo treatment for skin laxity of the abdomen.
* Subject's score on the skin laxity scale for skin on the abdomen is 1 (mild) or 2 (moderate).
* Subject agrees to maintain his/her weight (i.e., within 5%) by not making any major changes in diet, exercise or medication routine during the course of the study.
* Subject agrees to refrain from taking any medication(s) or supplements(s), whether prescription or OTC, or undergo any procedures indicated for weight loss, or for fat reduction or improving the appearance of the skin in the abdominal area (e.g. liposuction, ultrasound therapy) for the duration of participation in the clinical study.
* Willing to have research photos taken of treatment areas.
* Understands, and is able and willing to comply with all study visits, treatments and evaluations schedules and requirements.
* Females are at least 9 months post-partum.
* Females are post-menopausal, surgically sterilized, or using a medically accepted form of birth control for at least 3 months prior to the study and agree to continue to do so for the duration of study participation.

Exclusion Criteria:

* Skin laxity resulting from genetic disorders, including but not limited to Ehlers-Danlos Syndrome.
* History of undergoing a fat reduction procedure (e.g., liposuction, bariatric surgery, abdominoplasty).
* Botulinum toxin or other aesthetic drug injections within the abdomen area within the past 6 months.
* History of any major prior surgery in the abdominal area
* Implanted medical prostheses (such as clips, pins or plates) in or adjacent to the area of intended treatment.
* Active implanted device such as a pacemaker, defibrillator, or drug delivery system.
* Any clinical and significant dermatological skin condition(s) in the intended abdominal treatment area, such as skin infections or rashes, extensive scarring, psoriasis, etc..
* Tattoo or former tattoo at the treatment area.
* Current moderate to heavy tobacco use, defined as smoking 10 or more cigarettes per day (or equivalent use of other nicotine-containing products such as cigars, pipes, chewing tobacco, or e-cigarettes) within the past 6 months
* History of chronic drug or alcohol abuse.
* Pregnant or intending to become pregnant in the next 6 months.
* Currently enrolled in a clinical study of an unapproved investigational drug or device.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of accurately identified subject pre- and post-treatment photographs by at least two of the three Blinded Independent Evaluators. | 12 weeks
  Reviewers will be blinded to post-treatment (12 weeks) vs. baseline untreated area. The order in which images will be presented will be randomized. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form. Success is defined as at least 2 of the 3 blinded evaluators correctly identifying a subject's pre-treatment and post-treatment (study endpoint) photographs for 80% or more of subjects.

SECONDARY OUTCOMES:
Global Aesthetic Improvement Scale | 12 weeks
  The Global Aesthetic Improvement Scale (GAIS) is a widely used subjective qualitative assessment tool in clinical trials to evaluate the effectiveness of aesthetic interventions from before to after treatment using a five-point scale ranging from "3: very much improved" to "-1: worse," that enables investigators to provide a standardized evaluation of treatment outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Cesar A. Lara M.D. Weight Loss & Wellness, Dunedin, Florida, United States

IPD SHARING:
Plan to Share IPD: No